CLINICAL TRIAL: NCT03525171
Title: Comparison Between Euglycemic Hyperinsulinemic Clamp and Surrogate Indexes of Insulin Sensitivity in Children With Growth Hormone Deficiency.
Brief Title: Evalutation of Insulin Sensitivity Through Hyperinsulinemic Clamp in Children With GH Deficiency
Acronym: clamp-GHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Carla Giordano, Principa Investigator, University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: clamp-GHD
Record Dates: First submitted 2017-10-25; First posted 2018-05-15 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Intervention Model Description: We prospectively studied 23 prepubertal children with GH deficiency treated with GH for at least 12 months and 12 healthy subjects with short stature, matched for age and pubertal status
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GHD children (Active Comparator): 23 prepubertal children with isolated GHD consecutively admitted to the Section of Endocrinology of the University of Palermo during treated with GH for at least 12 months underwent full metabolic evaluation including euglycemic hyperinsulinemic clamp
  Interventions: Diagnostic Test: euglycemic hyperinsulinemic clamp
- controls (Placebo Comparator): 12 prepubertal healthy subjects with short stature recruited among children referred for assessment of short stature as a control group at baseline underwent full metabolic evaluation including euglycemic hyperinsulinemic clamp
  Interventions: Diagnostic Test: euglycemic hyperinsulinemic clamp

INTERVENTIONS:
Diagnostic Test: euglycemic hyperinsulinemic clamp — In addition to auxological and baseline biochemical parameters, we performed the clamp to evaluate insulin sensitivity (M-value) at baseline (GHD group and controls) and after 12 months of GH treatment (GHD group).

SUMMARY:
Data about the impact of growth hormone treatment on insulin sensitivity in children are quite controversial, due to the different surrogate indexes that have been used, like Homa-IR, QUICKI, ISI-Matsuda or adipokine levels.

The investigators aimed to evaluate insulin sensitivity through the euglycemic hyperinsulinemic clamp, considered the gold standard technique, in children affected by growth hormone deficiency and to compare the M-value with the most commonly used surrogate indexes of insulin sensitivity.

DETAILED DESCRIPTION:
The investigators aimed of this study was to use the hyperinsulinemic clamp to evaluate the impact of GH treatment on insulin-stimulated glucose utilization (M-value) in a group of children affected by GH deficiency and to compare the clamp-derived index with the most commonly used surrogate indexes of insulin sensitivity.

In all patients the auxological and metabolic evaluation was performed at baseline and after 12 months of GH treatment, while in controls these evaluations were only performed at baseline. In all children the investigators measured body height, body mass index (BMI) and waist circumference (WC). A blood sample was drawn after an overnight fast for the measurement of glucose, insulin, Hemoglobin A1c (HbA1c) and IGF-I. This sample served as the baseline for the oral glucose tolerance test (OGTT). Blood samples were collected every 30 min for 120 min for glucose and insulin measurements. As surrogate estimates of insulin sensitivity the investigators used the insulin sensitivity index, a composite index derived from the OGTT and validated by Matsuda and DeFronzo (ISI-Matsuda). On a different day, as a gold standard measurement of insulin sensitivity the investigators performed the euglycemic hyperinsulinemic clamp. As other insulin sensitivity markers, the serum levels of adiponectin and resistin after an overnight fast were also measured.

ELIGIBILITY:
Inclusion Criteria:

* Isolated idiopathic GH deficiency diagnosed by the auxological and biochemical criteria of the GH Research Society in prepubertal children
* Prepubertal children

Exclusion Criteria:

* Children with multiple hormone deficiency
* Children receiving other hormonal replacement treatment
* Pubertal children

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Change in insulin sensitivity in GHD children | baseline and after 12 months of GH treatment
  insulin sensitivity degree derived from clamp was calculates and compared with other indexes of insulin sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology - University of Palermo, Palermo, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data available on request, to expand and contine the study